CLINICAL TRIAL: NCT04630171
Title: Does the VerTouch Device Improve Insertion Site Identification for Lumbar Neuraxial Procedures When Compared to Palpation or Ultrasound Guided Site Selection? A Prospective Randomized Controlled Trial
Brief Title: VerTouch Device: A Prospective Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Intuitap (Unknown)
Responsible Party: Principal Investigator, Mahesh Vaidyanathan, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU00213282
Record Dates: First submitted 2020-11-12; First posted 2020-11-16 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Pain
Keywords: Pregnancy; Neuraxial Anesthesia; Therapeutic Lumbar Puncture; Ultrasound; Labor epidural; Spinal Procedure
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant
Masking Description: Participant will be blinded to what procedure will be used to identify lumbar landmarks.
  All devices will be in the room with the operator of the devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Group 1: VerTouch for labor epidural or spinal anesthesia procedure (Experimental): VerTouch utilized for identification of site for labor epidural or spinal anesthesia procedure in women requesting labor analgesia.
  Interventions: Device: Group #1: VerTouch utilized for identification of site for labor epidural or spinal anesthesia procedure
- Group 2: Ultrasound (US) for labor epidural or spinal anesthesia procedure (Active Comparator): Ultrasound (US) utilized for identification of site for labor epidural or spinal anesthesia procedure in women requesting labor analgesia.
  Interventions: Device: Group #2: Ultrasound (US) utilized for identification of site for labor epidural or spinal anesthesia procedure
- Group 3: Control group, palpation for labor epidural or spinal anesthesia procedure (Active Comparator): Control group, palpation utilized for identification of site for labor epidural or spinal anesthesia procedure in women requesting labor analgesia.
  Interventions: Other: Group #3: Control group, palpation utilized for identification of site for labor epidural or spinal anesthesia procedure

INTERVENTIONS:
Device: Group #1: VerTouch utilized for identification of site for labor epidural or spinal anesthesia procedure — Group #1: VerTouch utilized for identification of site for labor epidural or spinal anesthesia procedure for women requesting labor analgesia
  Other Names: Group 1
  Arms: Group 1: VerTouch for labor epidural or spinal anesthesia procedure
Device: Group #2: Ultrasound (US) utilized for identification of site for labor epidural or spinal anesthesia procedure — Group #2: Ultrasound (US) utilized for identification of site for labor epidural or spinal anesthesia procedure for women requesting labor analgesia
  Other Names: Group 2
  Arms: Group 2: Ultrasound (US) for labor epidural or spinal anesthesia procedure
Other: Group #3: Control group, palpation utilized for identification of site for labor epidural or spinal anesthesia procedure — Control group, palpation utilized for identification of site for labor epidural or spinal anesthesia procedure for women requesting labor analgesia
  Other Names: Group 3
  Arms: Group 3: Control group, palpation for labor epidural or spinal anesthesia procedure

SUMMARY:
This study will compare the VerTouch device to palpation and ultrasound (US) techniques used to identifying the anatomic landmarks and optimal location for neuraxial access. This trial of the VerTouch device will be compared to the gold standard of palpation and the commonly cited US techniques.

DETAILED DESCRIPTION:
Thousands of neuraxial procedures are completed daily with over 12,000 done at Prentice Women's hospital last year. These procedures are not without difficulty and complication. The gold standard of palpation and blind advancement of the needle toward the spine can result in multiple insertions of the needle into the skin and redirections of the trajectory of that needle after insertion to avoid the bones of the spine protecting the spinal column. These insertions and redirections are not only time consuming while the patient is in an uncommon position, but they also cause dis-comfort and possibly lasting pain days after the procedure. In addition to the patient dynamics, when anatomical or positioning issues result in difficult neuraxial procedures the common teaching is to attempt US guided access. Unfortunately, not many proceduralist are trained in this modality and the additional materials needed to perform the procedure with US take time to gather and further prolong the procedure. Additionally, though the cost of US technology is getting more reasonable, it is still rather expensive and a barrier to utilization by many facilities around the country and the world. Often, after many attempts, the proceduralist accepts failure of the procedure and refers the patient to the interventional radiology (IR) or pain medicine specialist for completion of the procedure using radiation to visualize the spine. Note, this is not an option for pregnant women who are not eligible for radiation due to fetal concerns.

The VerTouch device offers a non-invasive, untethered, and non-radiation producing device that allows for the visualization of the underlying structures of the spine to determine ideal needle placement for neuraxial procedures. The output on the screen can also be visualized by other providers or senior proceduralist for assistance with best course of action for the procedure. The device does not cause discomfort to the patient and does not require any additional materials to be functional.

Study participants will be recruited from Prentice Women's Hospital (Northwestern Medicine). Pregnant patients tend to be healthy and without comorbidities, and the anesthesiologists who perform the neuraxial procedure tend to have significant experience. Non-pregnant patients tend to require neuraxial access for diagnostic or therapeutic purposes (i.e. not for the relief of labor pains), and therefore have comorbidities.

Labor & Delivery: Participants will be randomized to one of the three arms (palpation, US, or VerTouch).

This study has the potential to show that the VerTouch is more effective than palpation and as effective as US at defining the location for neuraxial procedure initiation and eventual success.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years old and above
* Undergoing a neuraxial procedure

Exclusion Criteria:

* Non English speaking
* Plastic allergy
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Vaidyanathan, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital and Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 3: Control Group, Palpation for Labor Epidural or Spinal Anesthesia Procedure | Group 2: Ultrasound (US) for Labor Epidural or Spinal Anesthesia Procedure | Group 1: VerTouch for Labor Epidural or Spinal Anesthesia Procedure
Started | 28 | 26 | 32
Completed | 28 | 26 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: VerTouch for Labor Epidural or Spinal Anesthesia Procedure | Group 2: Ultrasound (US) for Labor Epidural or Spinal Anesthesia Procedure | Group 3: Control Group, Palpation for Labor Epidural or Spinal Anesthesia Procedure | Total
Number analyzed (Participants) | 32 | 26 | 28 | 86
Age, Continuous [Mean (Full Range); unit: Years] | 34.4 [22 to 42] | 34.3 [24 to 41] | 34.6 [21 to 42] | 34.3 [21 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 28 | 86
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 6
  White | 25 | 20 | 20 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 4 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 2 | 6 | 4 | 12
  Non-Hispanic | 30 | 19 | 23 | 72
  Not reported | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 26 | 28 | 86
BMI = Weight (kg) / Height (m)² [Mean (Full Range); unit: kg/m^2] | 29.32 [22.06 to 44.7] | 31.6 [22.36 to 41.79] | 31.12 [24.64 to 39.27] | 30.58 [22.06 to 44.7]
Height (in) [Mean (Full Range); unit: Inches] | 65.09 [58 to 70] | 64.69 [59 to 68] | 64.51 [59 to 67] | 64.8 [58 to 70]
Weight (Kilograms) [Mean (Full Range); unit: Kilograms] | 80.01 [58.8 to 110.9] | 85.2 [66.8 to 129.9] | 83.5 [62.1 to 102.8] | 84.04 [58.8 to 129.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Redirections of the Needle
Description: Primary endpoint is the number of redirections of the needle
Time Frame: End of procedure
Measure: Mean (Standard Deviation); unit: Number of redirections of needle
Arm/Group | Group 1: VerTouch for Labor Epidural or Spinal Anesthesia Procedure | Group 2: Ultrasound (US) for Labor Epidural or Spinal Anesthesia Procedure | Group 3: Control Group, Palpation for Labor Epidural or Spinal Anesthesia Procedure
Number analyzed (Participants) | 32 | 26 | 28
Number of redirections of needle | .72 (.9) | 2.81 (3.7) | 2.35 (3.9)

2. Secondary Outcome: Number of Reinsertions of the Needle
Description: Secondary endpoint is the number of reinsertions of the needle.
Time Frame: 24 hours.
Measure: Mean (Standard Deviation); unit: Number of needle insertions
Arm/Group | Group 1: VerTouch for Labor Epidural or Spinal Anesthesia Procedure | Group 2: Ultrasound (US) for Labor Epidural or Spinal Anesthesia Procedure | Group 3: Control Group, Palpation for Labor Epidural or Spinal Anesthesia Procedure
Number analyzed (Participants) | 32 | 26 | 28
Number of needle insertions | .11 (.3) | .96 (1.5) | .5 (1.0)

3. Secondary Outcome: Total Procedure Time
Description: Total neuraxial procedure time in minutes
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: VerTouch for Labor Epidural or Spinal Anesthesia Procedure | Group 2: Ultrasound (US) for Labor Epidural or Spinal Anesthesia Procedure | Group 3: Control Group, Palpation for Labor Epidural or Spinal Anesthesia Procedure
Number analyzed (Participants) | 32 | 26 | 28
Minutes | 8.66 (2.6) | 9.81 (4.1) | 7.88 (3.1)

ADVERSE EVENTS:
Time Frame: 24 hours after the neuraxial procedure.
Arm/Group | Group 1: VerTouch for Labor Epidural or Spinal Anesthesia Procedure | Group 2: Ultrasound (US) for Labor Epidural or Spinal Anesthesia Procedure | Group 3: Control Group, Palpation for Labor Epidural or Spinal Anesthesia Procedure
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 0/32 | 0/26 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT04630171/Prot_SAP_000.pdf